CLINICAL TRIAL: NCT03907072
Title: A Randomized, Double-blind, Placebo-controlled, Efficacy and Safety Study of WVE-210201 With Open-label Extension in Ambulatory Patients With Duchenne Muscular Dystrophy (DYSTANCE 51)
Brief Title: Efficacy and Safety Study of WVE-210201 (Suvodirsen) With Open-label Extension in Ambulatory Patients With Duchenne Muscular Dystrophy
Acronym: DYSTANCE 51
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Wave Life Sciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WVE-DMDX51-003
Record Dates: First submitted 2019-04-05; First posted 2019-04-08 (Actual); Results first posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-04

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- WVE-210201 (3 mg/kg) (Experimental): Weekly IV administrations of WVE-210210 at 3 mg/kg
  Interventions: Drug: WVE-210201 (suvodirsen)
- WVE-210201 (4.5 mg/kg) (Experimental): Weekly IV administrations of WVE-210210 at 4.5 mg/kg
  Interventions: Drug: WVE-210201 (suvodirsen)
- Placebo (Placebo Comparator): Weekly IV administrations of phosphate buffered saline solution visually identical in appearance to WVE-21021
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: WVE-210201 (suvodirsen) — WVE-210201 is a stereopure antisense oligonucleotide (ASO)
  Arms: WVE-210201 (3 mg/kg); WVE-210201 (4.5 mg/kg)
Drug: Placebo — Buffered saline solution
  Arms: Placebo

SUMMARY:
This is a Phase 2/3, multicenter, randomized, double-blind, placebo-controlled study with an open-label extension period to evaluate the safety and efficacy of WVE-210201 (suvodirsen) in ambulatory male pediatric patients with Duchenne muscular dystrophy (DMD) amenable to exon 51 skipping intervention (DYSTANCE 51)

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of DMD based on clinical phenotype with increased serum creatine kinase
2. Documented mutation in the Dystrophin gene associated with DMD that is amenable to exon 51 skipping
3. Ambulatory male, able to walk independently for at least 10 meters in 10 seconds or less at the time of Screening visit (performed as part of the NSAA)
4. Stable pulmonary and cardiac function, as measured by:

   1. Reproducible percent predicted forced vital capacity (FVC) ≥50%
   2. Left ventricular ejection fraction (LVEF) >55% in patients <10 years of age and >45% in patients ≥10 years of age, as measured (and documented) by echocardiogram
5. Currently on a stable corticosteroid therapy regimen, defined as initiation of systemic corticosteroid therapy occurred ≥6 months prior to Screening, and no changes in dosing ≤3 months prior to Screening visit

Exclusion Criteria:

1. Cardiac insufficiency:

   1. Severe cardiomyopathy that, in the opinion of the Investigator, prohibits participation in this study; however, cardiomyopathy that is managed by angiotensin-converting-enzyme (ACE) inhibitors or beta blockers is acceptable provided the patient meets the LVEF inclusion criterion
   2. Any other evidence of clinically significant structural or functional heart abnormality
   3. A cardiac troponin I value > 0.2 ng/mL
2. Need for daytime mechanical or non-invasive ventilation OR anticipated need for daytime mechanical or non-invasive ventilation within the next year, in the opinion of the Investigator. Nighttime non-invasive ventilation is permitted
3. Received prior treatment with drisapersen or with an investigational peptide-conjugated phosphorodiamidate morpholino oligomer (PPMO)
4. Received prior treatment with gene therapy for DMD
5. Received treatment with ataluren or eteplirsen within the 14 weeks prior to the planned Baseline biopsy collection
6. Received any investigational drug within 3 months or 5 half-lives, whichever is longer, prior to the planned Baseline biopsy collection

Ages: 5 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2020-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Panzara, MD, MPH, Study Director — Wave Life Sciences
Locations (22):
- United States (6):
  - Yale University, New Haven, Connecticut
  - Rare Disease Research, LLC., Atlanta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - University of Massachusetts, Worcester, Massachusetts
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Belgium (3):
  - Institut de Myologie, Liège, Liege
  - UZ Gent, Ghent
  - Universitaire Ziekenhuizen Leuven, Leuven
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - London Health Sciences Centre - Hospital, London, Ontario
- Fakultni Nemocnice v Motole, Prague, Czechia
- France (3):
  - Hôpitaux Universitaires de Strasbourg, Strasbourg, Bas-Rhin
  - Hôpital Des Enfants, Toulouse, Haute-Garonne
  - Hopital Armand Trosseau, Paris
- Italy (4):
  - Ospedale Pediatrico Bambino Gesù, Rome, Lazio
  - U.O.C di Neurologia e Malattie Neuromuscolari Centro Clinico Nemo Sud, Messina
  - Ospedale San Reffaele Via Olgettina, 60, Milan
  - Fondazione Policlinico Universitario A Gemelli, Roma
- Drottning Silvias Barn Och Ungdomssjukhus, Gothenburg, Sweden
- United Kingdom (2):
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Great Ormond Street Hospital (GOSH), London

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | WVE-210201 (3 mg/kg) | WVE-210201 (4.5 mg/kg) | Placebo
Started | 2 | 2 | 2
Completed | 0 | 0 | 0
Not Completed | 2 | 2 | 2
Not completed — Study Terminated by Sponsor | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | WVE-210201 (3 mg/kg) | WVE-210201 (4.5 mg/kg) | Placebo | Total
Number analyzed (Participants) | 2 | 2 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 2 | 6
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 6.5 [5 to 8] | 9 [8 to 10] | 7 [5 to 9] | 7.5 [5 to 10]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 2 | 2 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 2 | 2 | 5
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Sweden | 0 | 1 | 0 | 1
  Belgium | 1 | 0 | 0 | 1
  Italy | 0 | 0 | 2 | 2
  France | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Dystrophin Level (% Normal Dystrophin)
Description: US/other regions (as applicable)
Time Frame: Day 1 to Week 12, Week 22, or Week 46
Population: No statistical analysis has been performed due to early study termination
Arm/Group | WVE-210201 (3 mg/kg) | WVE-210201 (4.5 mg/kg) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Change From Baseline in North Star Ambulatory Assessment (NSAA)
Description: European Union (EU)/other regions (as applicable)
Time Frame: Day 1 through Week 48
Population: No statistical analysis has been performed due to early study termination.
Arm/Group | WVE-210201 (3 mg/kg) | WVE-210201 (4.5 mg/kg) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in North Star Ambulatory Assessment (NSAA)
Description: US/other regions (as applicable)
Time Frame: Day 1 through Week 48
Population: No statistical analysis has been performed due to early study termination.
Arm/Group | WVE-210201 (3 mg/kg) | WVE-210201 (4.5 mg/kg) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in Dystrophin Level (% Normal Dystrophin)
Description: European Union (EU)/other regions (as applicable)
Time Frame: Day 1 to Week 12, Week 22, or Week 46
Population: No statistical analysis has been performed due to early study termination.
Arm/Group | WVE-210201 (3 mg/kg) | WVE-210201 (4.5 mg/kg) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Change From Baseline in Upper Limb Proximal Strength
Time Frame: Day 1 through Week 48
Population: No statistical analysis has been performed due to early study termination.
Arm/Group | WVE-210201 (3 mg/kg) | WVE-210201 (4.5 mg/kg) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change From Baseline in 4-stair Climb
Time Frame: Day 1 through Week 48
Population: No statistical analysis has been performed due to early study termination.
Arm/Group | WVE-210201 (3 mg/kg) | WVE-210201 (4.5 mg/kg) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline in the 10-meter Walk/Run Test
Time Frame: Day 1 through Week 48
Population: No statistical analysis has been performed due to early study termination.
Arm/Group | WVE-210201 (3 mg/kg) | WVE-210201 (4.5 mg/kg) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline in Forced Vital Capacity
Time Frame: Day 1 through Week 48
Population: No statistical analysis has been performed due to early study termination.
Arm/Group | WVE-210201 (3 mg/kg) | WVE-210201 (4.5 mg/kg) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Change From Baseline in the 95th Percentile of Stride Velocity
Time Frame: Day 1 through Week 48
Population: No statistical analysis has been performed due to early study termination.
Arm/Group | WVE-210201 (3 mg/kg) | WVE-210201 (4.5 mg/kg) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Change From Baseline in NSAA
Description: Long-term evaluation, open label from Week 48 through Week 96
Time Frame: Day 1 through Week 96
Population: No statistical analysis has been performed due to early study termination.
Arm/Group | WVE-210201 (3 mg/kg) | WVE-210201 (4.5 mg/kg) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Study enrollment through early study termination by Sponsor (maximum of 11 weeks).
Arm/Group | WVE-210201 (3 mg/kg) | WVE-210201 (4.5 mg/kg) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WVE-210201 (3 mg/kg) (N=2) | WVE-210201 (4.5 mg/kg) (N=2) | Placebo (N=2)
Cardiac Disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WVE-210201 (3 mg/kg) (N=2) | WVE-210201 (4.5 mg/kg) (N=2) | Placebo (N=2)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (4) | 0 (0)
Pyrexia (General disorders) | 1 (3) | 2 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (4) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/72/NCT03907072/Prot_SAP_000.pdf